CLINICAL TRIAL: NCT03898583
Title: A Phase 1b, Randomised, Controlled, Assessor-blinded Proof of Principle Trial to Assess Safety, Tolerability and Pharmacodynamics Effects of Microarray Patches Containing Calcipotriol/Betamethasone Dipropionate in Descaled Skin of Adults With Chronic Plaque Psoriasis Over a 21-day Treatment Period
Brief Title: Clinical Trial to Assess Safety, Tolerability and the Pharmacodynamics Effect of Calcipotriol/Betamethasone Dipropionate in a New Administration Form in Subjects With Chronic Plaque Psoriasis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LP0120-1391
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; betamethasone-17,21-dipropionate; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison of all treatments
Who Masked: Investigator
Masking Description: The trial will be assessor-blinded with random assignment of the 2 microarray patches containing calcipotriol and betamethasone dipropionate, the vehicle (microarray patches without active substance) and the active comparator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microarray patch A (Experimental): 21 day treatment, once weekly, 3 applications in total, transdermal patch for cutaneous use
  Interventions: Drug: Microarray patch A
- Microarray patch B (Experimental): 21 day treatment, 3 times weekly, 9 applications in total, transdermal patch for cutaneous use
  Interventions: Drug: Microarray patch B
- Vehicle (Placebo Comparator): 21 day treatment, once weekly, 3 applications in total, transdermal patch for cutaneous use, no active substance
  Interventions: Drug: Placebo
- Daivobet (Active Comparator): 21 day treatment, paused on day 7, day 14 and day 21, Cutaneous use
  Interventions: Drug: Daivobet

INTERVENTIONS:
Drug: Microarray patch A — Microarray patch
  Other Names: Calcipotriol; Betamethasone dipropionate
  Arms: Microarray patch A
Drug: Microarray patch B — Microarray patch
  Other Names: Calcipotriol; Betamethasone dipropionate
  Arms: Microarray patch B
Drug: Placebo — Microarray patch vehicle
  Arms: Vehicle
Drug: Daivobet — Daivobet Gel
  Other Names: Calcipotriol; Betamethasone dipropionate
  Arms: Daivobet

SUMMARY:
To assess safety, tolerability and pharmacodynamics effect of treatment with microarray patches containing calcipotriol and betamethasone dipropionate.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with psoriasis vulgaris in a chronic stable phase and mild to moderate plaque(s) covering a sufficient area to allocate 4 test fields on up to 3 comparable plaques.
* Men and women aged 18-70 years (inclusive).
* Sufficient target lesion(s) must be present on the trunk or extremities (excluding palms/soles); psoriatic lesions on the knees or elbows are not to be used as target lesions.
* Plaques to be treated should have a comparable thickness of the EPB of the inflammatory infiltrate of at least 200 μm.
* Plaques to be treated should have no more than a 2-fold difference in infiltrate thickness between the test fields.
* Physical examination of skin must be without abnormal, clinical significant findings other than psoriasis vulgaris unless the investigator considers an abnormality to be irrelevant to the trial outcome.

Key Exclusion Criteria:

* Other skin disease noted on physical examination that is considered by the investigator to be relevant to the outcome of the trial.
* Subjects with acute psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica, pustular, exfoliative or inverse psoriasis.
* History of psoriasis that was unresponsive or poorly responsive to topical treatments.
* Topical antipsoriatics are not permitted on the same body area as plaques to be treated during the 4 weeks before first treatment and during the trial.
* Systemic treatment with antipsoriatics e.g. corticosteroids, cytostatics, retinoids, dimethylfumarate, apremilast in the 3 months before first treatment and during the trial.
* Systemic treatment with biological treatments: rituximab within 12 months, ustekinumab or secukinumab within 6 months before first treatment and during the trial.
* Systemic treatment with biological treatments within 3 months before first treatment and during the trial.
* Systemic treatment with any other biological treatments within the period of 5 half-lives of the biological before first treatment and during the trial.
* UV-therapy or extensive exposure to UV radiation or sunlight within 4 weeks before first treatment and during the trial.
* Treatment with concomitant medication that may affect and provoke or aggravate psoriasis, unless on a stable dose for 3 months before trial medication initiation.
* Any other topical medication on the plaques to be treated during the trial.
* Clinically significant abnormal vital signs (blood pressure, and pulse) at screening (V1).
* History/symptoms of a clinically significant illness before first treatment (past 5 years) and during the trial that in the investigator's opinion may place the subject at risk.
* History/symptoms of a clinically significant illness before first treatment (past 5 years) and during the trial that in the investigator's opinion may influence the trial outcome.
* Other clinically significant abnormal laboratory results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Overall number of treatment-emergent adverse events. | First IMP application up to trial end (Day 50)
Number of treatment-emergent application site reactions, by treatment | First IMP application up to trial end (Day 50)
Change from baseline to Day 22 (EoT) in haematology parameters. | From baseline up to EoT (Day 22)
  RBC, WBC, haemoglobin, haematocrit, platelets, white cell differentials; measured in SI units.
Change from baseline to Day 22 (EoT) in clinical chemistry parameters. | From baseline to EoT (Day 22)
  Sodium, potassium, BUN, glucose, AST, ALT, gamma GT, AP, calcium, phosphate, albumin, total cholesterol, LDH, total protein, creatinine, total bilirubin; measured in SI units.
Change from baseline to Day 22 (EoT) in urinalysis parameters, single parameters only to be listed if deviation from usual urine dip test. | From baseline to EoT (Day 22)
  E.g., leukocytes, nitrite, pH, protein, glucose, ketones, urobilinogen, bilirubin, blood/haemoglobin, measured in SI units.
Number of subjects with abnormal clinically significant findings of physical examination at Day 22 (EoT). | EoT (Day 22)
  Evaluation of physical examination (areas skin, heart, lung, abdomen, basic neurological status, general examination of eyes, ears, nose, throat), overall evaluation, assessed by investigator as 'normal', 'abnormal not clinically significant', 'abnormal clinically significant'.
Change from baseline to Day 22 (EoT) in systolic and diastolic blood pressure. | From baseline to EoT (Day 22)
  Measured in mmHg.
Change from baseline to Day 22 (EoT) in pulse. | From baseline to EoT (Day 22)
  Measured in beats per minute.
Frequency counts of overall tolerability assessment of skin reactions at Day 8, Day 15, Day 22, Day 36 and Day 50. | From baseline up to trial end (Day 50)
  (Assessment performed by an investigator using a 4-point score ['0 = very good', '1 = good', '2 = moderate', '3 = poor']).

SECONDARY OUTCOMES:
Change from baseline (pre-dose at Day 1) to Day 22 (EoT) in psoriatic infiltrate thickness. | EoT (Day 22)
  (Assessed by measurement of the thickness of the Echo Poor Band [EPB] of the inflammatory infiltrate using 22-MHz sonography; measured in µm).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (2):
- Germany (2):
  - LEO Pharma investigational site, Berlin
  - LEO Pharma investigational site, Hamburg

IPD SHARING:
Plan to Share IPD: No